CLINICAL TRIAL: NCT04932317
Title: Oral Symptom Assessment Scale (OSAS): Validity and Reliability
Status: Completed | Type: Observational
Sponsor: Our Lady's Hospice and Care Services (Other)
Collaborators: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Prof Andrew Davies, Professor of Palliative Medicine, Our Lady's Hospice and Care Services
Other Study IDs: PM202166
Record Dates: First submitted 2021-03-30; First posted 2021-06-21 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Neoplasms
Keywords: Oral health; Oral care; Neoplasms; Palliative care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oral (mouth) symptoms are very common and often bothersome in patients with cancer. The best way to assess these symptoms is using a patient-rated symptom assessment scale. A new symptom assessment scale for oral symptoms has been developed and already tested in patients. The purpose of this study is to test the scale again to make sure it is reliable and accurate.

DETAILED DESCRIPTION:
Oral health is multifaceted and includes an individual's ability to speak, eat as well as to convey emotion without pain, embarrassment or discomfort. Oral health contributes to an individual's general well-being.

Poor oral health in patients with advanced cancer can be associated with negative impacts on an individual's quality of life in terms of psychological and emotional distress (e.g. avoiding social interactions due to embarrassment) and physical distress (e.g. pain associated with mucositis). As well as this certain problems can be associated indirectly with mortality in patients with advanced cancer e.g. oral infection leading to systemic infection.

In patients with advanced cancer oral symptoms are common, often multiple and of high-impact. Routine screening for oral symptoms should be undertaken in all patients with advanced cancer in conjunction with regular examination of the oral cavity to ensure correct diagnosis and adequate treatment.

A novel oral symptom assessment scale (OSAS) was designed and developed to measure the frequency, severity and distress (or bother) of twenty oral symptoms in patients with advanced cancer. This initial observational study provided provisional validation of the new assessment tool.

This study aims to further investigate the reliability and validity of this novel oral symptom assessment tool in patients with advanced cancer. Test-retesting will occur in patients deemed clinically stable. Test- retesting will be undertaken to measure reliability on two occasions 24-48 hours apart. Recruited patients will be asked to fill in the OSAS as well as the EORTC QLQ- C30 and EORTC QLQ-OH15 (a validated quality of life assessment with an oral health module) which will provide criterion (concurrent) validity.

ELIGIBILITY:
Inclusion Criteria

* Any cancer diagnosis
* Age ≥ 18 years old
* Able to understand and speak English
* Signed witnessed consent form
* In the 'Stable' clinical phase

Exclusion Criteria

* In the judgement of the Palliative Care physician, study participation is not appropriate
* Unable to complete the study assessments in entirety i.e. in full at Time 1 ( 0 hours) and at Time 2 (24 hours later)
* In the 'Unstable', 'Deteriorating' or 'Terminal' clinical phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer admitted to a specialist palliative care in-patient unit
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
To measure the reliability of the oral symptom assessment scale (i.e assess if any change) | Measured at Time 1 ( Time 1 = 0 hours ) and Time 2 (Time = 24 hours later)
  The oral symptom assessment scale is a twenty-question patient-reported symptom assessment scale. Participants are asked to rate how often ( rarely, occasionally, frequently, almost constantly), the severity (slight, moderate, severe, very severe) and distress or bother ( not at all, a little bit, somewhat, quite a bit, very much) of any of these twenty oral symptoms during the past week.
To measure the concurrent validity of the OSAS against the EORTC QLQ-OH15 | Measured at Time 1 ( Time = 0 hours)
  The European Organisation for Research and Treatment of Cancer Quality of Life of cancer patients questionnaire is a patient-reported outcomes evaluation of quality of life in cancer patients and the European Organisation of Research and Treatment of Cancer Quality of Life Oral Health questionnaire is an oral health quality of life module. The former consists of thirty questions assessing five functions, nine symptoms and global health status/quality of life. The EORTC QLQ OH-15 module consists of one multi-item scale to assess oral health quality of life and five single items to assess sore mouth, sticky saliva, sensitivity, dentures and information.All of the scales and single-item measures range in score from 0 to 100.A high score for the functional scale and single item represents a high level of functioning, this is, a low level of symptomatology or problems. A high score for the symptom items represents a high level of symptomatology or problems.
To measure ease of use | Measured at Time 1 ( Time = 0 hours)
  Participants will be asked to fill in an ease of use questionnaire at Time point 1. The two questions will be yes or no answers ( 1. Did you think the OSAS was easy to complete? 2. Did you think the EORTC QLQ C30 and EORTC QLQ OH15 was easy to complete?)

OTHER OUTCOMES:
Ease of answering questionnaire | At Time 1 only ( Time 1 = 0 hours)
  Participants will be asked about how easy the questionnaires are to answer i.e the two questions posed are : "Did you think Questionnaire 1 (OSAS) was easy to complete?" Answer: Yes or No and " Did you think Questionnaire 2 (EORTC QLQ-C30 and EORTC QLQ-OH15) was easy to complete?" Answer: Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Davies, MB FRCP, Principal Investigator — Our Lady's Hospice, Harold's Cross, Dublin 6W Ireland
Locations (1):
- Our Lady's Hospice and Care Services, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glick M, Williams DM, Kleinman DV, Vujicic M, Watt RG, Weyant RJ. A new definition for oral health developed by the FDI World Dental Federation opens the door to a universal definition of oral health. J Am Dent Assoc. 2016 Dec;147(12):915-917. doi: 10.1016/j.adaj.2016.10.001. No abstract available. PMID 27886668
- [Background] Hjermstad MJ, Bergenmar M, Fisher SE, Montel S, Nicolatou-Galitis O, Raber-Durlacher J, Singer S, Verdonck-de Leeuw I, Weis J, Yarom N, Herlofson BB. The EORTC QLQ-OH17: a supplementary module to the EORTC QLQ-C30 for assessment of oral health and quality of life in cancer patients. Eur J Cancer. 2012 Sep;48(14):2203-11. doi: 10.1016/j.ejca.2012.04.003. Epub 2012 May 8. PMID 22572480
- [Background] Davies, A. 2010. Oral care in advanced cancer patients. In: Davies A.N. and Epstein J.B. (eds) Oral Complications of Cancer and Its Management. Oxford University Press, Oxford, pp279-289
- [Background] Davies A, Buchanan A, Todd J, Gregory A, Batsari KM. Oral symptoms in patients with advanced cancer: an observational study using a novel oral symptom assessment scale. Support Care Cancer. 2021 Aug;29(8):4357-4364. doi: 10.1007/s00520-020-05903-1. Epub 2021 Jan 8. PMID 33416995
- [Background] Shah S, Davies AN. Re: medical records vs. patient self-rating. J Pain Symptom Manage. 2001 Oct;22(4):805-6. doi: 10.1016/s0885-3924(01)00348-7. No abstract available. PMID 11596613
- [Background] Aktas A, Walsh D, Kirkova J. The psychometric properties of cancer multisymptom assessment instruments: a clinical review. Support Care Cancer. 2015 Jul;23(7):2189-202. doi: 10.1007/s00520-015-2732-7. Epub 2015 Apr 19. PMID 25894883
- [Background] Hjermstad MJ, Bergenmar M, Bjordal K, Fisher SE, Hofmeister D, Montel S, Nicolatou-Galitis O, Pinto M, Raber-Durlacher J, Singer S, Tomaszewska IM, Tomaszewski KA, Verdonck-de Leeuw I, Yarom N, Winstanley JB, Herlofson BB; EORTC QoL Group. International field testing of the psychometric properties of an EORTC quality of life module for oral health: the EORTC QLQ-OH15. Support Care Cancer. 2016 Sep;24(9):3915-24. doi: 10.1007/s00520-016-3216-0. Epub 2016 Apr 25. PMID 27113466
- [Background] Paiva CE, Barroso EM, Carneseca EC, de Padua Souza C, Dos Santos FT, Mendoza Lopez RV, Ribeiro Paiva SB. A critical analysis of test-retest reliability in instrument validation studies of cancer patients under palliative care: a systematic review. BMC Med Res Methodol. 2014 Jan 21;14:8. doi: 10.1186/1471-2288-14-8. PMID 24447633
- [Background] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Background] Smith, M . Palliative care casemix - stage 2 development: a national classification for any site of care. 8th national casemix conference, Sydney, NSW, Australia, 16-18 September 1996. Canberra, ACT, Australia: Commonwealth Department of Human Services and Health.
- [Background] Koo TK, Li MY. A Guideline of Selecting and Reporting Intraclass Correlation Coefficients for Reliability Research. J Chiropr Med. 2016 Jun;15(2):155-63. doi: 10.1016/j.jcm.2016.02.012. Epub 2016 Mar 31. PMID 27330520
- [Background] Arifin, W.N. 2018. A Web-based Sample Size Calculator for Reliability Studies. Educational Resources. https://pdfs.semanticscholar.org/0bf5/ddcc23d91a941fa0bacf992de1f970e33a1c.pdf